CLINICAL TRIAL: NCT07323329
Title: Growth Hormone and Dehydroepiandrosterone Effect on Poor Ovarian Reserve Patients During in Vitro Fertilization
Brief Title: Growth Hormone and Dehydroepiandrosterone Role in Vitro Fertilization
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Lecturer of Clinical Pharmacy, Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/01092024/Ragab
Record Dates: First submitted 2025-12-17; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Infertility; Infertility (IVF Patients)
Keywords: Growth hormone; Infertility; IVF patients; Ovarian reserve
MeSH Terms: conditions — Infertility | interventions — Human Growth Hormone; Folic Acid; Dehydroepiandrosterone; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Somatropin group (Experimental): Somatropin (4IU for 1 month) 1 S.C injection every 3 days for at least 1 month plus, folic acid 400mcg/day
  Interventions: Drug: Somatropin (4IU for 1 month) plus, folic acid 400 mcg per day.
- dehydroepiandrosterone (Experimental): dehydroepiandrosterone 50 mg twice per day for 12 weeks plus folic acid 400mcg per day
  Interventions: Drug: DHEA plus folic acid 400mcg per day
- Standard care (Active Comparator): Patients will receive standard care will receive folic acid 400 mcg per day
  Interventions: Dietary Supplement: control group

INTERVENTIONS:
Drug: Somatropin (4IU for 1 month) plus, folic acid 400 mcg per day. — Patients will receive Somatropin (4IU for 1 month)1 S.C injection every 3 days for at least 1 month plus, folic acid 400 mcg per day.
  Arms: Somatropin group
Drug: DHEA plus folic acid 400mcg per day — Patients will receive DHEA 50 mg twice per day for 12 weeks plus folic acid 400mcg per day
  Arms: dehydroepiandrosterone
Dietary Supplement: control group — Patients will receive folic acid 400 mcg per day
  Arms: Standard care

SUMMARY:
The goal of this study is to evaluate the role of Somatropin and Dehydroepiandrosterone (DHEA) on ovarian reserve parameters and intracytoplasmic sperm injection (ICSI) outcome in poor ovarian responder.

The main question it aims to answer is:

Which intervention is more effective in increasing number and size of follicles? Participants will be followed 1 month before starting induction in growth hormone and 12 weeks for DHEA and through intracytoplasmic sperm injection (ICSI) cycle.

ELIGIBILITY:
Inclusion Criteria:

At least two of the following three criteria had to be present after maximal stimulation:

1. Advanced maternal age (>40 years) or any other risk factor for Poor Ovarian Response (POR).
2. ≤3 oocytes with a conventional stimulation protocol).
3. An abnormal ovarian reserve test [i.e. antral follicle count (AFC) less than 5-7 follicles or anti-Müllerian hormone (AMH) below 0.5-1.1 ng/ml].

Exclusion Criteria:

1. Any endocrine or metabolic disorder such as hyperprolactinemia, diabetes and thyroid dysfunction.
2. Any pelvic pathology such as hydrosalpinx, uterine anomaly.
3. Any male factor infertility such as Oligo-Astheno-Teratozoospermia (OAT) or azoospermia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 165 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
The number of mature oocyte | 12 weeks

SECONDARY OUTCOMES:
pregnancy rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casson PR, Lindsay MS, Pisarska MD, Carson SA, Buster JE. Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series. Hum Reprod. 2000 Oct;15(10):2129-32. doi: 10.1093/humrep/15.10.2129. PMID 11006185
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20231167/